CLINICAL TRIAL: NCT01704989
Title: A Randomised Controlled Trial to Compare the Clinical Effectiveness of Selective Laser Trabeculoplasty (SLT) Versus Topical Therapy in the Treatment of Pseudoexfoliative Glaucoma
Brief Title: The Laser in Pseudoexfoliation (LIP) Study
Acronym: LIP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not submit to the REB
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LIP-SLT-2012
Record Dates: First submitted 2012-09-18; First posted 2012-10-12 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2012-10

CONDITIONS: Glaucoma
Keywords: Glaucoma, SLT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser pathway (Active Comparator): Arm in which patients first randomised to receive SLT laser
  Interventions: Procedure: SLT Laser
- Topical therapy (Active Comparator): Arm in which patients first selected to receive drops (Prostagladin analogue as first-line)
  Interventions: Drug: Prostagladin

INTERVENTIONS:
Procedure: SLT Laser — At the first treatment, SLT treatment will be delivered to 360 degrees of trabecular meshwork. At the first escalation of treatment, the superior 180 degrees will be retreated. Twenty-five non-overlapping shots per quadrant will be used with a starting power of 0.8 mJ and increments of 0.1 mJ (titrated to avoid large bubbles) with standard other settings (400 nm spot size, 3 nanosecond duration) using a Latina single-mirror goniolens. The IOP will be checked 1 hour post treatment and five days of guttae acular tds will be administered to the treatment eye following treatment. After 2 treatments of SLT, the laser treated arm of the study will follow the same pathway as the medical treatment arm.
  Other Names: Slective Laser Trabeculoplasty (primary treatment)
  Arms: Laser pathway
Drug: Prostagladin — Treatment will be initiated with latanoprost 0.005%. At the first IOP check (1-2 months), if the IOP has not reached target IOP, a second line agent will be added (β-Blocker unless contraindicated). If target IOP is still not reached, a third agent will be considered (topical carbonic anhydrase inhibitor). Treatment may be switched, instead, at the discretion of the clinician if the reduction of IOP with an agent is deemed to be no different than the pre-treatment IOP. Surgical therapy will be considered if target IOP is not met, or there is high IOP (>35 mmHg) or advanced damage at presentation.
  Other Names: B-Blocker; Carbonic anydrase inhibitor
  Arms: Topical therapy

SUMMARY:
A number of large clinical trials have found pseudoexfoliation (PXF) to be a major risk factor for glaucoma progression and risk of blindness. It is estimated that PXF accounts for approximately a quarter of cases of open angle glaucoma in Nova Scotia, Canada, making this region an ideal setting for studying patients with this condition. Despite associated high morbidity, the treatment of pseudoexfoliative glaucoma remains suboptimal and a challenge for the clinician. Topical medical therapy is less effective than for primary open angle glaucoma and patients often require early surgical therapy, with associated risks. Selective laser trabeculoplasty (SLT) may be a safe and effective treatment for pseudoexfoliative glaucoma, although the evidence for this is presently lacking. The aim of the current study is to provide the first controlled-trial evidence for the effectiveness of SLT, compared to topical therapy, in the management of pseudoexfoliative glaucoma.

DETAILED DESCRIPTION:
Objectives:

The primary aim of this study is to compare the effectiveness, in terms of intraocular pressure (IOP) control, of SLT and topical medical therapy in the primary treatment of patients with high IOP secondary to PXF. The secondary aims of the study are:

1. To examine the relationship between the degree of angle pigmentation and reduction of IOP
2. To examine adverse effects from SLT treatment in patients with PXF
3. To compare IOP-lowering effects of SLT in patients with PXF to patients with POAG (in the LiGHT study, see structure below).

Study Population: All new patients with PXF who are naïve to treatment (and willing to participate) will be recruited after their first hospital consultation. Both eyes will be treated but only one eye per patient included in the analysis (eye with the higher presenting IOP).

Structure: The study design mirrors that of National Institute of Health (NIHR-) funded, the laser in glaucoma and ocular hypertension trial (LiGHT) in the UK and is a collaborative study between a Canadian Institute and Moorfields Eye Hospital in London. This is a single-study randomised (unmasked) control trial of a proposed treatment intervention (SLT) versus a standard treatment (topical therapy).

Summary of study design Patients will be randomised to one of 2 trial arms: 'laser-pathway' or 'medicine- pathway'. Following initial treatment, SLT patients will be followed up 1-2 weeks after treatment to check IOP and for potential side effects. The interval of subsequent follow-up visits (between 4 and 12 months) will be governed by the level of IOP in relation to the target IOP and the severity of glaucoma. Visual field testing (SITA standard, 24-2 test pattern) and imaging with the Hedidelberg Retina Tomograph (HRT III) will be performed at each visit. Target IOP will be set using the Canadian Glaucoma Society guidelines depending on the severity of glaucoma and the level of IOP. At subsequent visits, treatment will be escalated if the target IOP is not met or if there is evidence of progression.

Duration of study The study will last 3 years. One year will be allowed for recruitment of all study participants, so that a minimum follow-up of 2 years will be available.

All patients will have a medical history, gonioscopy, central corneal thickness (CCT) measurement, IOP measurement with Goldmann applanation tonometry and dilated fundoscopy at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of PXF material on the anterior chamber structures by slit lamp biomicroscopy.
* An open drainage angle with no irido-trabecular contact on non-indentation gonioscopy in primary position trabecular meshwork visible over 360 degrees.
* Ocular hypertension or glaucoma deemed to require treatment by the attending clinician.
* A decision to treat has been made by a Consultant Glaucoma Specialist.
* Age over 18 years and able to provide informed consent.

Exclusion Criteria:

* Advanced glaucoma as determined by EMGT criteria 1: visual field loss mean deviation worse than -12 dB in the better or -15 dB in the worse eye.
* Co-existing other secondary glaucoma (e.g. pigment dispersion syndrome, rubeosis etc) or angle closure glaucoma.
* History of retinal ischaemia, macular oedema or diabetic retinopathy.
* Age-related macular degeneration with neovascularisation or geographic atrophy and VA worse than 6/36.
* Any previous intra-ocular surgery, except uncomplicated phacoemulsification at least one year before.* Medically unfit for completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of drops (and surgical interventions) needed to reach target IOP. | Change in IOP at 6 months, 12 months and 2 years (from baseline).
Percentage success | At 6 months, 12 months and 2 years
  Proportion of patients in whom SLT (or mono medical therapy) alone achieved target IOP.

SECONDARY OUTCOMES:
Correlation of angle pigment grade with IOP reduction from SLT | 6 months, 12 months, 2 years
Comparison of percentage success and number of drops in current study with the equivalent results of patients with POAG in the LiGHT study | 1 year and 2 years
Number of progressing patients in each study arm (SLT or medical therapy) in terms of visual field loss and HRT. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo T Nicoela, MD, Principal Investigator — Capital District Health Authority/Dalhousie University
Locations (1):
- Eye Care Centre, VG Site, QEII, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114